CLINICAL TRIAL: NCT05682690
Title: Laparoscopic Eradication of Deep Endometriosis With Nerve-sparing Rectosigmoid Segmental Resection: a Comparative Retrospective Analysis (RSRES_NERVSP)
Brief Title: Laparoscopic Eradication of Deep Endometriosis With Nerve-sparing Rectosigmoid Segmental Resection (RSRES_NERVSP)
Acronym: RSRES_NERVSP
Status: Completed | Type: Observational
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-ZF
Record Dates: First submitted 2022-11-03; First posted 2023-01-12 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center, retrospective case-control study. All consecutive women who underwent classic and nerve-sparing segmental rectosigmoid resection between January 2005 and June 2022 will be included. In the majority of cases classic segmental rectosigmoid resection was done between January 2005 and December 2010. Nerve-sparing segmental rectosigmoid resection has been increasingly employed since January 2011 until now. Preoperative (anamnestic, physical objective, and ultrasonographic data), surgical and postoperative data of the patients included in this study will be analyzed. In particular, postoperative data will be obtained by analyzing reports of follow-up visits, which are routinely done at our institution at 1, 6, 12 months and then every year following the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* consecutive women who underwent classic and nerve-sparing segmental rectosigmoid resection between January 2005 and June 2022
* age more than 18 years.

Exclusion Criteria:

* diagnosis of other/concomitant preoperative and/or postoperative medical or surgical conditions altering pelvic organ function (i.e. multiple sclerosis, irritable bowel syndrome);
* age <18 years.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with rectosigmoid endometriosis who underwent classic or nerve-sparing segmental rectosigmoid resection between January 2005 and June 2022
Sampling Method: Non-Probability Sample
Enrollment: 3072 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Number of patients having intraoperative complications | During the surgical procedures
  Number of patients having intraoperative complications evaluated by surgical data stored in the hospital medical electronic register
Number of patients having short-term postoperative complications | 3 months after the surgical procedures
  Number of patients having short-term postoperative complications evaluated by clinical data stored in the hospital medical electronic register at the follow-up visits
Number of patients having middle-term postoperative complications | 6 months after the surgical procedures
  Number of patients having short-term postoperative complications evaluated by clinical data stored in the hospital medical electronic register at the follow-up visits
Number of patients having long-term postoperative complications | 12 months after the surgical procedures
  Number of patients having short-term postoperative complications evaluated by clinical data stored in the hospital medical electronic register at the follow-up visits

SECONDARY OUTCOMES:
Intraoperative blood loss (ml) | During the surgical procedures
  Intraoperative blood loss (ml) evaluated by surgical data stored in the hospital medical electronic register
Number of patients having an intraoperative laparotomic conversion | During the surgical procedures
  Intraoperative blood loss (ml) evaluated by surgical data stored in the hospital medical electronic register
Operative time (min) | During the surgical procedures
  Operative time (min) evaluated by surgical data stored in the hospital medical electronic register
Number of patients undergoing a concomitant additional surgical procedure | During the surgical procedures
  Number of patients undergoing a concomitant additional surgical procedure evaluated by surgical data stored in the hospital medical electronic register

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Ceccaroni, Principal Investigator — IRCCS Sacro Cuore Don Calabria
Locations (1):
- IRCCS Sacro Cuore Don Calabria di Negrar, Negrar, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ceccaroni M, Ceccarello M, Raimondo I, Roviglione G, Clarizia R, Bruni F, Mautone D, Manzone M, Facci E, Rettore L, Rossini R, Bertocchi E, Barugola G, Ruffo G, Barra F. "A Space Odyssey" on Laparoscopic Segmental Rectosigmoid Resection for Deep Endometriosis: A Seventeen-year Retrospective Analysis of Outcomes and Postoperative Complications among 3050 Patients Treated in a Referral Center. J Minim Invasive Gynecol. 2023 Aug;30(8):652-664. doi: 10.1016/j.jmig.2023.04.005. Epub 2023 Apr 26. PMID 37116746